CLINICAL TRIAL: NCT03925948
Title: Health Literacy Enhanced Intervention for Inner-city African Americans With Uncontrolled Diabetes: A Pilot Study
Brief Title: Health Literacy Intervention for African Americans With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Brancati Center for the Advancement of Community Care (Unknown); Center for Community Innovation and Scholarship at the Johns Hopkins University (Unknown); East Baltimore Medical Center (Unknown); Shepherds Clinic (Unknown); John Hopkins Aftercare Clinic (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00061339
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Uncontrolled Diabetes
Keywords: Type 2 diabetes; African American; numeracy; self-management; glucose control
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The investigators used a single-arm pre- and post-test design for this pilot study in which the investigators assessed the feasibility, acceptability, and preliminary efficacy of the PLAN 4 Success-Diabetes in inner-city AAs in Baltimore, Maryland. Community-dwelling AAs were recruited via referrals from inner-city federally-qualified health clinics. Nineteen of 30 participants who completed the baseline survey received the study intervention which consisted of four-week health literacy training and disease knowledge education followed by two home visits and monthly phone counseling for over 6 months.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): This is a one arm study with all participants enrolled into this arm.
  Interventions: Behavioral: PLAN 4 Success-Diabetes

INTERVENTIONS:
Behavioral: PLAN 4 Success-Diabetes — The study intervention-PLAN 4 Success-Diabetes-consisted of four 1 to 1 ½-hour weekly health literacy training and disease knowledge education sessions for four weeks (4 in-person sessions), followed by two home visits and monthly phone counseling for over 6 months (5 phone sessions). The intervention is theory-driven and builds on von Wagner's model to incorporate key elements such as health literacy, disease knowledge, and self-efficacy for better glucose outcomes.

SUMMARY:
Disparities in diagnosis and control of type 2 diabetes mellitus are most evident in African Americans (AAs) with lower socioeconomic status. Health literacy is an important predictor of adequate self-management and control of diabetes. The purpose of this pilot study was to test the feasibility and preliminary efficacy of a health literacy-enhanced diabetes intervention -Prevention through Lifestyle intervention And Numeracy (PLAN) 4 Success-Diabetes, in inner-city, low-income AAs with uncontrolled diabetes. To evaluate the feasibility, acceptability, and preliminary efficacy of the intervention, the investigators conducted a pilot study with 24-week follow-up. The investigators that participation in the PLAN 4 Success-diabetes intervention would be associated with a reduction in glucose outcomes and improvements in psychosocial variables.

ELIGIBILITY:
Inclusion Criteria:

* African Americans residing in Baltimore, Maryland
* had uncontrolled diabetes (defined as HbA1C>7%)

Exclusion Criteria:

* Unable to give informed consent
* Physical or mental health conditions that could limit active participation in the study (e.g., blindness in both eyes, severe immobility, psychiatric diseases)
* Hematological condition that would affect HbA1C assay, e.g., hemolytic anemia, sickle cell anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-05-06 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Health literacy as assessed by Literacy Assessment in Diabetes (LAD). | baseline; 12 and 24 weeks
  The Literacy Assessment in Diabetes (LAD) has high reliability and validity indices. The items on the LAD are scored as correct/incorrect, with total possible scores ranging from 0 to 60. Higher scores indicated higher health literacy levels.
Change in Health literacy as assessed by the Newest Vital Sign | baseline; 12 and 24 weeks
  The Newest Vital Sign consists of four items and measures numeracy. After reviewing a nutrition label, participants are asked to answer questions based on some calculation of the nutritional information (e.g., fat, sodium) presented on the label. Total possible scores range from 0 to 4, with one point assigned for each correct response.

SECONDARY OUTCOMES:
Change in Diabetes knowledge measured with the validated Diabetes Knowledge Test | baseline; 12 and 24 weeks
  The Diabetes Knowledge Test assesses diabetes knowledge, medications, diet, and management with questions such as "What effect will an infection most likely have on blood glucose." Correct responses are given a score of one.
Change in Diabetes self-efficacy measured with Stanford Diabetes Self-Efficacy scale | baseline; 12 and 24 weeks
  The Stanford Diabetes Self-Efficacy scale assesses participant's efficacy in managing diabetes and maintaining healthy lifestyles. The scale asks how confident participants are in managing different tasks such as eating meals every 4 to 5 hours every day or breakfast every day measured on a Likert scale of 0 "not at all confident" to 10 "totally confident." Participant scores are the means across all items in the instrument.

OTHER OUTCOMES:
Change in Diabetes self-care index | baseline; 12 and 24 weeks
  This index included seven questions on smoking, alcohol consumption, meal planning, consumption of high fat foods, consumption of high sugar foods, consumption of sodium, and medium or high intensity exercise. These questions were coded into dichotomous responses with participation in healthy behaviors coded as "1" and active participation in negative health behaviors coded as "0". A summary score for the index could range 0-7 and higher scores indicate better self-care.
Change in Social support as assessed by modified Medical Outcomes Study-Social Support Survey (mMOS-SS) | baseline; 12 and 24 weeks
  mMOS-SS is a shorter version (10 items) of the Medical Outcomes Study-Social Support Survey (MOS-SS) which includes 19 items. The original version was used to measure social support in community dwelling chronically ill persons. mMOS-SS covers emotional and instrumental domains of social support with strong evidence of reliability and validity. Example items include: "How often is someone available to take you to the doctor if you need it" or "How often is someone available who understands your problems?" Response options are from all of the time (5 point) to none of the time (1 point) with higher scores indicating higher levels of social support (total score range=10 to 50).
Change in Depression status as assessed by the Patient Health Questionnaire (PHQ)-9 | baseline; 12 and 24 weeks
  The Patient Health Questionnaire (PHQ)-9 addresses the severity of depressive symptoms based on the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV). The PHQ-9 has 9 items scored from 0 (not at all) to 3 (nearly every day) with total scores ranging from 0 to 27. Individuals are asked whether any symptom(s) have been experienced over the past 2 weeks. Evidence of reliability, validity, sensitivity, and specificity has been reported in community samples.
Change in Quality of Life as assessed by the EuroQol Quality of Life scale | baseline; 12 and 24 weeks
  It contains the EQ-5D-3L that provides a single index of health status. The EQ-5D-3L assess five domains; mobility, self-care, usual activities, pain/discomfort and anxiety/depressions. Responses show if participants do not have difficulty, have some problems or have severe difficulty within the domains. Summary scores for the sample were created across each of the five items (range 0-2) with higher scores indicating better quality of life. A component of this scale is the EuroQol visual analogue scale (EQ-VAS) which participants can use a number from 0-100 to identify participant's health state.

CONTACTS AND LOCATIONS:
Overall Officials: Hae-Ra Han, PhD, RN, Principal Investigator — Johns Hopkins University
Locations (1):
- Wald Community Nursing Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] von Wagner C, Steptoe A, Wolf MS, Wardle J. Health literacy and health actions: a review and a framework from health psychology. Health Educ Behav. 2009 Oct;36(5):860-77. doi: 10.1177/1090198108322819. Epub 2008 Aug 26. PMID 18728119
- [Derived] Han HR, Nkimbeng M, Ajomagberin O, Grunstra K, Sharps P, Renda S, Maruthur N. Health literacy enhanced intervention for inner-city African Americans with uncontrolled diabetes: a pilot study. Pilot Feasibility Stud. 2019 Aug 8;5:99. doi: 10.1186/s40814-019-0484-8. eCollection 2019. PMID 31410294